CLINICAL TRIAL: NCT03826524
Title: CanROC Epinephrine Dose: Optimal Versus Standard Evaluation Trial (CanROC EpiDOSE Trial)
Brief Title: Epinephrine Dose: Optimal Versus Standard Evaluation Trial
Acronym: EpiDOSE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EpiDOSE Protocol Version 3.0
Record Dates: First submitted 2018-11-07; First posted 2019-02-01 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Sudden Cardiac Arrest; Ventricular Fibrillation; Ventricular Tachycardia-Pulseless
Keywords: out-of-hospital cardiac arrest; sudden cardiac arrest; epinephrine; randomized controlled trial
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Death, Sudden, Cardiac; Ventricular Fibrillation | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose Epinephrine (Active Comparator): Epinephrine up to 2mg total
  Interventions: Drug: Epinephrine
- Standard Dose Epinephrine (Active Comparator): Epinephrine up to 6mg total
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Epinephrine — Epinephrine 1mg 1:10000 (10cc) per dose
  Other Names: Adrenaline

SUMMARY:
The objective of this randomized controlled trial is to evaluate the effectiveness of a low cumulative dose of epinephrine compared to a standard cumulative dose of epinephrine during resuscitation from ventricular fibrillation (VF) or ventricular tachycardia (VT) in adult out-of-hospital cardiac arrest (OHCA) patients.

DETAILED DESCRIPTION:
This study is designed as a prospective, multicentre, single-blinded randomized controlled trial (RCT) where eligible OHCA patients are randomized to receive a low cumulative dose of epinephrine (low dose epinephrine, up to 2mg total) or a standard cumulative dose of epinephrine (standard dose epinephrine, up to 6mg total) in a 1:1 fashion.

Eligible OHCA patients will be treated by paramedics who will initiate cardiopulmonary resuscitation (CPR) and the delivery of defibrillation shocks per paramedic agencies' treatment protocols. After one defibrillation and when feasible, paramedics will establish peripheral intravenous (IV) access, and patients will be randomly allocated to either the low dose or standard dose treatment arm. Epinephrine doses (according to treatment assignment) will be administered every 3-5 minutes, based on current guidelines and paramedic protocols, until the first return of spontaneous circulation (ROSC) is achieved or if resuscitation has been terminated by the base hospital physician. Other medications (e.g. antiarrhythmics, magnesium, beta blockers) and interventions (e.g. intubation) may be interposed as required. Follow-up will take place using a combination of administrative databases (e.g. the Discharge Abstract Database and the National Ambulatory Care Reporting System) and telephone interviews.

This RCT will evaluate a fundamental change in the treatment of OHCA. The investigators hypothesize that a low cumulative dose of epinephrine will improve patient survival to hospital discharge compared to a standard cumulative dose of epinephrine. Please feel free to contact epidose@unityhealth.to for further information.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest treated by paramedics
* Initial recorded cardiac rhythm of VF or pulseless VT, or, AED shock on first analysis administered or witnessed by EMS (paramedic or fire)
* Established intravenous vascular access

Exclusion Criteria:

* Known or apparent age <18 years
* Initial recorded cardiac rhythm of VF or pulseless VT, or, AED shock on first analysis administered or confirmed by paramedics
* Cardiac arrest due to an obvious non-cardiac primary cause (e.g. blunt or penetrating trauma, exsanguination, burns, drug overdose, drowning, anaphylaxis, sudden asphyxiation, etc.)
* Administration of intramuscular, endotracheal tube, or intraosseous epinephrine
* Prisoners or persons in police custody
* Known allergy or sensitivity to epinephrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3790 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Survival to hospital discharge | Through study completion (up to 5 years)
  Individuals discharged alive from hospital

SECONDARY OUTCOMES:
Return of spontaneous circulation in out-of-hospital setting | Through study completion (up to 5 years)
  Return of spontaneous circulation in the field
Survival to emergency department arrival | Through study completion (up to 5 years)
  Individuals alive upon arrival to a hospital emergency department
Survival to admission with death prior to discharge | Through study completion (up to 5 years)
  Individuals alive upon hospital admission who die in-hospital before being discharged
Survival to discharge outside of a long-term healthcare facility e.g. nursing home | Through study completion (up to 5 years)
  Individuals discharged alive from hospital to a care facility
Modified Rankin Scale (mRS) score | 12+/-3 months
  Assessment of neurological function, scores range from 0 to 6 where higher scores indicate worse neurological function (0=no symptoms, 6=dead)
Health Utility Index-3 (HUI-3) score | 12+/-3 months
  Assessment of quality of life, scores range from -0.36 to 1 where higher scores indicate better quality life (negative scores=a state worse than being dead, 0=dead, 1=perfect health)
Hospital Anxiety and Depression Scale score | 12+/-3 months
  Assessment of quality of life, scores range from 0 to 21 where higher scores indicate more anxiety/depression
Length of stay in hospital | Through study completion (up to 5 years)
  Length of time an individual remained in-hospital (length in days)
Length of stay in critical care unit | Through study completion (up to 5 years)
  Length of time an individual remained in a crucial care unit (length in days)
Survival post-arrest | Up to 5 years
  Survival following hospital discharge, up to 5 years
Recurrent cardiac arrest(s) | Up to 5 years
  Number of cardiac arrests following the index arrest
ICD implant post-arrest | Up to 5 years
  Whether an implantable cardioverter defibrillator was implanted post-arrest
Cardiovascular re-hospitalization(s) | Up to 5 years
  Number of cardiovascular re-hospitalizations
All-cause re-hospitalizations(s) | Up to 5 years
  Number of re-hospitalizations for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dorian, MD, MSc, Principal Investigator — Unity Health Toronto; Steve Lin, MD, MSc, Principal Investigator — Unity Health Toronto
Locations (8):
- Canada (8):
  - British Columbia Emergency Health Services (BCEHS), Victoria, British Columbia
  - Peel Regional Paramedic Services, Brampton, Ontario
  - Middlesex-London Paramedic Service, London, Ontario
  - Halton Region Paramedic Services, Oakville, Ontario
  - Ottawa Paramedic Services, Ottawa, Ontario
  - Superior North Emergency Medical Services, Thunder Bay, Ontario
  - Essex-Windsor Emergency Health Services, Windsor, Ontario
  - Medavie Health Services West, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No